CLINICAL TRIAL: NCT01647997
Title: Effects of an Acute Administration of Bacterial Endotoxin on Whole Body and Regional Lactate Metabolism in Healthy Male Volunteers
Brief Title: Lactate Metabolism After an Endotoxin Challenge in Healthy Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne (Other)
Collaborators: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Luc Tappy, MD, Professor of Physiology, University of Lausanne
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Lsne-128/01
Record Dates: First submitted 2012-07-17; First posted 2012-07-24 (Estimated); Last update posted 2012-07-24 (Estimated); Status verified 2012-07

CONDITIONS: Sepsis
Keywords: bacterial lipopolysaccharides; hyperlactatemia; muscle lactate
MeSH Terms: conditions — Sepsis; Hyperlactatemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- study 1a (Experimental): whole body lactate production after bacterial endotoxin challenge
  Interventions: Other: bacterial endotoxin challenge
- study 1b (No Intervention): basal whole body lactate production
- study 2a (Experimental): muscle lactate concentration after bacterial endotoxin challenge
  Interventions: Other: bacterial endotoxin challenge
- study 2b (No Intervention): basal muscle lactate concentrations

INTERVENTIONS:
Other: bacterial endotoxin challenge — iv administration of 2ng/kg bacterial endotoxin
  Arms: study 1a; study 2a

SUMMARY:
Sepsis is characterized by hyperlactatemia, the severity of which is proportionate with sepsis severity. The pathophysiological mechanisms (increased lactate production vs decreased lactate utilization; tissues involved in sepsis-induced lactate production) remain largely unknown.

In this study, the investigators will assess whole body and regional metabolism in healthy young male subjects on two occasions, once after administration of an intravenous bacterial endotoxin challenge, and once without intervention.

In one group of subjects, whole body lactate metabolism will be measured over 10 hours after the endotoxin challenge

* Energy expenditure and net substrate oxidation rates (indirect calorimetry)
* Lactate kinetics (measured by means of a continuous, exogenous sodium lactate infusion)
* Glucose kinetics (measured with 6,6 d2 glucose)
* Hemodynamic parameters and body temperature
* Blood clinical chemistry In one group of subjects, whole body lactate metabolism will be measured over 10 hours after the endotoxin challenge
* Energy expenditure and net substrate oxidation rates (indirect calorimetry)
* Lactate kinetics (measured by means of a continuous, exogenous sodium lactate infusion)
* Glucose kinetics (measured with 6,6 d2 glucose)
* Hemodynamic parameters and body temperature
* Blood clinical chemistry

In a second group of subjects, regional muscle lactate metabolism will be measured over 10 hours after the endotoxin challenge by means of muscle microdialysis

ELIGIBILITY:
Inclusion Criteria:

* gender male
* body mass index (BMI) < 25 kg/m2
* absence of known disease

Exclusion Criteria:

* any known pathology
* abnormal cardio-pulmonary and hemodynamic status
* electrocardiographic alterations
* history of allergy
* current medications
* drug abuse
* consumption of more than 20g/day alcohol

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2002-04; Primary Completion 2004-03 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Whole body lactate production | single bacterial endotoxin administration; measurements over 6.5 hours following administration
  Whole body lactate clearance will be measured by measuring the increase in blood lactate at steady state during a conrtinuous exogenous sodium lactate infusion.
  Lactate production will be calculated as the product of lactate clearance times per-infusion blood lactate concentration
skeletal muscle lactate concentration | single bacterial endotoxin administration; measurements over 6.5 hours following administration
  interstitial muscle measured by means of in vivo microdialysis ; calculation of muscle-blood lactate gradient

SECONDARY OUTCOMES:
whole body energy expenditure | single bacterial endotoxin administration; measurements over 6.5 hours following administration
  open circuit indirect calorimetry (hood)
body temperature | single bacterial endotoxin administration; measurements over 6.5 hours following administration

CONTACTS AND LOCATIONS:
Overall Officials: René Chiolero, MD, Principal Investigator — Centre Hospitalier Universitaire Vaudois
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Derived] Michaeli B, Martinez A, Revelly JP, Cayeux MC, Chiolero RL, Tappy L, Berger MM. Effects of endotoxin on lactate metabolism in humans. Crit Care. 2012 Jul 27;16(4):R139. doi: 10.1186/cc11444. PMID 22839504